# Trial of Rucaparib in Patients With Metastatic Hormone-Sensitive Prostate Cancer Harboring Germline DNA Repair Gene Mutations

NCT03413995

3/31/2022

Date: March 31, 2022

Principal Investigator: Mark Markowski M.D. Ph.D.

Application No.: IRB00156514

NCT03413995

If appropriate for this study, a scanned copy of the signed consent form should be uploaded to the participant's Epic/EMR record.

Patient I.D. plate

# RESEARCH PARTICIPANT INFORMED CONSENT AND PRIVACY AUTHORIZATION FORM

Protocol Title: Phase II <u>Trial of Rucaparib in Patients with Metastatic and Non-</u>

**Metastatic Hormone-Sensitive Prostate Cancer Harboring DNA** 

**Repair Gene Mutations (TRIUMPH)** 

**Application No.:** IRB00156514

**Sponsor:** Clovis Oncology

Principal Investigator: Mark C. Markowski M.D., Ph.D.

Johns Hopkins Sidney Kimmel Comprehensive Cancer Center

401 North Broadway Baltimore, MD 21231 Phone: 410 955-8893 Fax: 410 955-8587

# 1. What you should know about this study:

- You are being asked to join a research study. This consent form explains the research study and your part in it. Please read it carefully and take as much time as you need. Ask your study doctor or the study team to explain any words or information that you do not understand.
- You are a volunteer. If you join the study, you can change your mind later. There will be no penalty or loss of benefits if you decide to quit the study.
- During the study, we will tell you if we learn any new information that might affect whether you wish to continue to participate.
- If we think your participation in this study may affect your clinical care, information about your study participation will be included in your medical record, which is used throughout Johns Hopkins. Doctors outside of Johns Hopkins may not have access to this information. You can ask the research team to send this information to any of your doctors.
- When Johns Hopkins is used in this consent form, it includes The Johns Hopkins University, The
  Johns Hopkins Hospital, Johns Hopkins Bayview Medical Center, Howard County General Hospital,
  Johns Hopkins Community Physicians, Suburban Hospital, Sibley Memorial Hospital and All
  Children's Hospital.
- Biospecimens will be collected in this study. Biospecimens may include any of the following: blood, tissue, saliva, urine, bone marrow, cells, etc. Most biospecimens contain DNA, which is the genetic code for each person.

Date: March 31, 2022

Principal Investigator: Mark Markowski M.D. Ph.D.

Application No.: IRB00156514

• A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

• If you would like to review the information for this study, or a summary of the results, ask the study team doctor for the ClinicalTrials.gov study registration number.

## 2. Why is this research being done?

This aim of this research is to find out if the study drug rucaparib lowers prostate-specific antigen (PSA) levels in men with recurrence of prostate cancer that has not yet been treated with androgen deprivation therapy (also referred to as a biochemical recurrence [if there is no evidence of cancer on staging imaging] or metastatic hormone sensitive prostate cancer [if cancer is evident on imaging]) and who have a mutation in a gene involved in repairing DNA damage. The research will also examine if rucaparib is safe in individuals with recurrent prostate cancer.

Prior research studies have shown that drugs like rucaparib can be of benefit to patients with advanced metastatic prostate cancer who are resistant to androgen deprivation therapy AND who carry a mutation in a DNA repair gene. We are studying if rucaparib will be effective for these patients earlier in their treatment course (for example, prior to the start of medicines that lower testosterone levels).

It is unknown whether rucaparib will have the same benefit in men with metastatic or biochemically recurrent prostate cancer carrying a mutation in a DNA repair gene, prior to the use of medicines that lower testosterone levels. Medicines that lower testosterone levels (also known as androgen deprivation therapy) is a Food and Drug Administration (FDA) approved therapy for metastatic prostate cancer and results in patients living longer. It may also be used in patients with biochemically recurrent prostate cancer in certain circumstances.

Participants in this research study will be refusing life-prolonging therapy. Medicines that lower testosterone levels (androgen deprivation therapy +/- docetaxel +/- abiraterone) will not be given to participants on this study.

Participants will remain eligible to receive androgen deprivation therapy after completing or withdrawing from this study.

Rucaparib tablets are approved by the FDA for the treatment of metastatic ovarian cancer that has progressed after at least 2 lines of prior chemotherapy, for patients with certain known DNA mutations. Rucaparib is also FDA- approved for use in metastatic prostate cancer that have become resistant to testosterone based therapies such as androgen deprivation therapy. The FDA is allowing the use of rucaparib in this research study.

All participants who enroll in the study will have the same procedures and receive the same study drug (rucaparib).

Men 18 years or older with metastatic prostate cancer, who have a mutation in a gene that affects repair of DNA damage and normal testosterone levels, may join the study.

#### How many people will be in this study?

Up to 30 participants are expected to enroll in this study. About 20 of these participants are expected to be enrolled at Johns Hopkins.

Date: March 31, 2022

Principal Investigator: Mark Markowski M.D. Ph.D.

Application No.: IRB00156514

# 3. What will happen if you join this study?

If you agree to be in this study, we will ask you to do the following things:

#### **Screening Period:**

There will be a screening period to see if you can participate in the study. During the screening period the following procedures will be performed:

- The study team will ask you questions about your medical history and health and review your medical record.
- A physical examination and vital signs (body temperature, blood pressure, pulse, respiratory rate, weight).
- Eastern Cooperative Oncology Group (ECOG) performance status score: This is a scale used to assess how your cancer is progressing, and how your cancer affects your daily living abilities.
- Review of other medications you are currently taking.
- Collection of a blood sample (about 3 tablespoons of blood) for laboratory tests which measure your blood chemistry, including kidney and liver function, count your red and white blood cells and platelets. Lab test to measure how long it takes your blood to clot.
- Collection of urine sample for routine analysis.
- Electrocardiogram (ECG): This test gives a picture of the electrical action of your heart.
- CT scan and bone scan (if these have not been performed in the past 8 weeks). Computed tomography (CT) scan or magnetic resonance imaging (MRI) of the known areas of disease. These pictures will allow your doctor to monitor your disease before, during and after you receive the study drugs. In addition, bone scans will be completed to measure your disease
- If you are eligible for the study and choose to participate, you will be scheduled for a biopsy of your cancer, which is required prior to the start of rucaparib.
  - O Bone biopsies are optional in this study. If you have tumor only in your bones, you have the option to decline the biopsy.
- Will you give permission to take part in the screening tumor biopsy of your bone?

| YES $\square$ | |
|---------------|--------------------------|
| | Signature of Participant |
| No 🗆 | |
| | Signature of Participant |

Date: March 31, 2022

Principal Investigator: Mark Markowski M.D. Ph.D.

Application No.: IRB00156514

| ) | If no, will y surgery? | ou give permission to obtain pathology slides from your previous prostatectomy |
|---|---|---|
| | YES □ | Signature of Participant |
| | NO 🗆 | Signature of Participant |

There are many different gene defects that can affect DNA repair. These genetic defects can be inherited or just be isolated to your tumor. To be able to participate on this study, you must have had prior genetic testing confirming the presence of a genetic alteration that can be inherited (called a germline mutation).

You will not be screened for inheritable genetic alterations as part of this study. If you have not been tested or do not have an inheritable genetic mutation in a gene that affects DNA repair, you are not eligible for this study.

If you qualify to continue to participate in the study based on the results of the screening visit tests and procedures, you will be scheduled for a clinic visit after which you will start on the rucaparib regimen.

All participants who enroll in the study will have the same procedures and receive the same study drug (rucaparib).

#### **Study Drug Administration Period:**

If you are found to be eligible to continue to participate in the study, you will return to the clinic to begin taking the study drugs. You will take two doses of study drug at the same time each day, morning and evening, about 12 hours apart, with one glass of water and with or without food. The tablets should be swallowed whole and not chewed, crushed, dissolved or divided.

If vomiting occurs shortly after the study drug tablets are swallowed, the dose should only be replaced if all of the intact tablets can be seen and counted. Should you miss a scheduled dose for whatever reason (such as forgetting to take the tablets or vomiting), you will be allowed to take the scheduled dose up to a maximum of 2 hours after that scheduled dose time. If greater than 2 hours after the scheduled dose time, the missed dose is not to be taken and you should take your next dose at the next scheduled time.

You will visit the study doctor as instructed. Each study drug cycle is about 4 weeks. The study doctor or staff will discuss with you when and on which days to report to the clinic.

Date: March 31, 2022

Principal Investigator: Mark Markowski M.D. Ph.D.

Application No.: IRB00156514

#### **During Cycles (Every 4 weeks)**

You will return to the clinic every 4 weeks. At each visit, the following tests and procedures will be performed:

- Review of any changes in your health and medications since your last visit.
- You will be asked about the symptoms you are having from your disease and side effects you
  may be experiencing.
- Measurement of your weight and vital signs.
- An evaluation of your ability to carry out daily activities will be performed.
- A physical examination.
- Collection of a blood sample (about 2 tablespoons of blood) for laboratory tests which measure your blood chemistry, including kidney and liver function, count your red and white blood cells and platelets.

#### **Every 3 months or 6 months:**

You will have a CT scan and bone scan every 3 months if you have metastatic disease and every 6 months if you do not have metastatic disease while you are enrolled in the study, as well as a CT and bone scan at the end of the study (if it has been at least 1 month since your last CT and bone scan).

#### The following tests will be done for research:

• Collection of a blood sample (about 1 tablespoon) for research at screening and at the time of disease worsening (progression).

## Change to Every 3 month Clinic Visits after more than 12 months of study drug:

Once you have been on the study for 12 months, you will return to the clinic every 3 months (12 weeks) for your study visits. At each visit, the following tests and procedures will be performed:

- Review of any changes in your health and medications since your last visit.
- You will be asked about the symptoms you are having from your disease and side effects you may be experiencing.
- Measurement of your weight and vital signs.
- An evaluation of your ability to carry out daily activities will be performed.
- A physical examination.
- Collection of a blood sample (about 2 tablespoons of blood) for laboratory tests which measure your blood chemistry, including kidney and liver function, count your red and white blood cells and platelets.

Date: March 31, 2022

Principal Investigator: Mark Markowski M.D. Ph.D.

Application No.: IRB00156514

#### **Optional tumor biopsy:**

We would like your permission to perform a second tumor biopsy after 12 weeks of receiving rucaparib. This procedure is optional. If you refuse to have a biopsy, this will not affect your participation on this study nor will it affect your future care.

Will you give permission to take part in this optional tumor biopsy after 12 weeks of rucaparib?

| YES 🗆 | Signature of Participant |
|-------|--------------------------|
| No □ | Signature of Participant |

#### End of Study Drug Regimen Visit/28-Day Follow-up Visit

If you complete all of the study drug regimen/intervention cycles or if you are withdrawn from the study at any time, you will come in for an end of study drug regimen visit 28 days after your last dose of study drug to have the following procedures done:

- Review of any changes in your health and medications since your last visit.
- Measurement of your weight and vital signs.
- An evaluation of your ability to carry out daily activities will be performed.
- A physical examination.
- Collection of a blood sample (about 2 tablespoons of blood) for laboratory tests which measure your blood chemistry, including kidney and liver function, count your red and white blood cells and platelets.
- Imaging tests: CT or MRI of the abdomen and pelvis, CT or MRI of the chest (or chest x-ray), and bone scan, as determined by the study doctor.

The procedures and visits in this clinical trial are different from the standard treatments. If you choose to join the study, there are more frequent clinic visits (every month instead of every 3 months), more frequent blood tests (monthly, then every month instead of every 3-6 months), and receiving rucaparib instead of standard treatments. The standard treatments are medicines that lower testosterone with the addition of chemotherapy in certain patients. You will not be receiving an FDA approved medication that has been shown in clinical studies to make patients with your type of cancer live longer.

The results from all study tests (blood tests, CT and bone scans) will be given to you and be available to your physicians. Genetic counseling (discussing of what the tests may mean for your health and the health of any family members who may also have the same genetic changes) will be available to you at your request.

Date: March 31, 2022

Principal Investigator: Mark Markowski M.D. Ph.D.

Application No.: IRB00156514

#### Request to collect and store biospecimens for future research

As part of this research study, we would like to ask you to let us store your biospecimens and health information for future research. This research could involve other diseases and involve research tools such as gene sequencing or creation of cell lines. These samples may also be distributed to other researchers, but they will not contain any information that could be used to identify you. You may limit the future use of any banked samples by contacting the study doctor.

The research may involve research tools such as gene sequencing or the creation of cell lines.

- Gene sequencing of your DNA provides researchers with the code to your genetic material.
- Cell lines are living tissue samples that can be grown in a laboratory. A cell line can provide an unlimited supply of cells in the future without requiring more samples from you. Each cell contains your complete DNA.

The Genetic Information Nondiscrimination Act (GINA) may help protect you from health insurance or health-related employment discrimination based on genetic information.

The law provides that health insurance companies and group health plans

- may not ask for genetic information from this research and
- may not use genetic information when making decision about eligibility or premiums

The law will not stop health insurance companies from using genetic information to decide whether to pay claims. The law does not apply to other types of insurance (such as life, disability or long-term care).

Despite the GINA protections and the best efforts of the research team to protect your information, you may still be at risk if information about you were to become known to people outside of this study.

The study doctor can provide you with additional information if you have questions. Also, further information about our use of your biospecimens can be found in this consent document under the heading *What happens to Data and Biospecimens that are collected in the study?* 

Will you allow us to store the biospecimens we collect for this study for use in future research?

| YES 🗆 | |
|-------|--------------------------|
| | Signature of Participant |
| No 🗆 | |
| | Signature of Participant |

Date: March 31, 2022

Principal Investigator: Mark Markowski M.D. Ph.D.

Application No.: IRB00156514

#### **Incidental Findings**

The imaging you are having as part of this research study will be reviewed by a qualified person just as it would be if you were having the imaging as part of your routine medical care.

There is a possibility that while reviewing your imaging we may see an abnormality that we did not expect to see in this study. This is what is called an "incidental finding."

We will let you know if we see such an incidental finding. Depending on the type of incidental finding, we may contact you by mail or by phone. In the case of a potential serious emergency, someone may go to your home.

A qualified person (usually a member of the research team) will talk to you if there is an incidental finding. You do not have an option to decline information about an incidental finding.

If you want, we will give information about this incidental finding to your primary doctor or we will refer you to an appropriate doctor for further evaluation.

- An incidental finding may cause you to feel anxious.
- Since an incidental finding will be part of your medical record, it may affect your current or future life or health insurance coverage. This risk will vary depending on the type of insurance plan involved.
- The costs for any care that will be needed to diagnose or treat an incidental finding would not be paid for by this research study. These costs would be your responsibility.

## How long will you be in the study?

We anticipate that most participants will be on the study for about 12 months. Some participants may be a part of the study for a shorter time period and some may be for a longer time period.

# 4. What are the risks or discomforts of the study?

It is important that you tell the study staff about any other medicines, vitamins, nutritional or herbal supplements you are taking before and during the study. It is possible that your study drug could affect your other medication and there are certain medications that you will not be allowed to take with the study drug during the study, including other anti-cancer therapies and certain vaccines. Your study doctor will provide you with a list of medications that you must avoid while you are taking your study drug, so it is important to consult your study doctor before taking anything new.

Side effects can be mild, moderate or severe (these are explained below).

- Mild: You are aware of the side effect but it doesn't really bother you
- Moderate: You need to take some sort of action (like painkillers for a headache)
- Severe: The side effect stops you doing what you normally would be doing

Rucaparib has been associated with the following laboratory findings and/or clinical symptoms, generally of mild or moderate severity and generally not requiring treatment to be stopped.

You may experience none, some or all of the side effects listed below.

#### Very common side effects (occur in 10% or more of patients):

- Nausea or vomiting (feeling sick or actually being sick): If required, you will be offered medication to control these symptoms.
- Fatigue: Including asthenia (feeling tired, weary, exhausted, lack of or loss of energy, weakness).

Date: March 31, 2022

Principal Investigator: Mark Markowski M.D. Ph.D.

Application No.: IRB00156514

• Low blood counts (red blood cells, white blood cells, and platelets). Sometimes fever occurs with the low blood counts. These low blood count effects may be more likely to occur after multiple cycles of treatment.

**Anemia:** The number of red cells in your blood may decrease, which may cause shortness of breath and in some instances may require blood transfusions (when you are given new blood or blood-based products from a donor). Low red blood cell count may make you feel tired or dizzy. If you feel dizzy while taking rucaparib, you should avoid potentially hazardous tasks such as driving or operating machinery.

- o **Neutropenia:** A low white blood cell count puts you at higher risk for bacterial or viral infections. Having a high temperature or fever while your white blood cell count is low is a medical emergency and you must proceed to the nearest emergency room as soon as possible.
- o **Thrombocytopenia:** The number of platelets (another type of cell) in your blood may decrease which could lead to bleeding events. Symptoms include but are not limited to easy bruising, prolonged bleeding from cuts, blood in stools or urine, or nose bleeding.
- A low phosphate level in your blood. Usually there are no symptoms but if the levels are critically low, you may notice trouble breathing, confusion, muscle weakness, and/or irritability.
- Increase in cholesterol: If required, you will be offered medication to lower your cholesterol.
- Changes in kidney and liver function blood tests. These changes will be evaluated by your study doctor along with any in the context of other side effects that you are experiencing as well as other test results
  - o Increase in AST/ALT in your blood. These are enzymes produced by your liver. This will be monitored by the laboratory safety tests that will be done in this study because this does not normally have any symptoms. If necessary, you will be told to stop taking rucaparib until your AST/ALT values return to normal.
  - O Increase in creatinine in your blood: (A laboratory test to measure how well your kidney is functioning): This will be monitored by the laboratory safety tests that will be done in this study. The increase in creatinine observed in patients receiving rucaparib was mild and did not result in impaired kidney function. Your doctor will monitor your creatinine levels during the study and may decide if you need any further tests.
- Dysgeusia: Taste changes which may affect the way food normally tastes.
- Stomach-related effects such as constipation, vomiting, diarrhea, decreased appetite, stomach pain (epigastric pain), and indigestion.
- Dyspnea: Shortness of breath
- Dizziness: If required, you will be offered medication to control these symptoms.
- Photosensitivity:
  - o It is possible that rucaparib may make your skin and eyes more sensitive to sunlight. You should take all of the usual sun protection precautions when going outside. It is advised that you avoid excessive sun exposure, wear protective clothing (including wearing a hat and sunglasses), and use sunscreens regularly (sun protection factor 50 or greater).
- Fever sometimes can occur independent of a low blood count. If you experience an elevation of your temperature, please refer to your study doctor for fever management.
- Difficulty sleeping

#### Common side effects: (occur in 1 to less than 10% of patients):

• Rash<sup>a</sup>: which will appear as changes in your skin color (e.g. redness) and texture (e.g. bumps, blisters, peeling). Some rashes may be itchy, painful, or cause no symptoms at all. This can vary in severity from mild to severe.

Date: March 31, 2022

Principal Investigator: Mark Markowski M.D. Ph.D.

Application No.: IRB00156514

• **Pruritis**<sup>a</sup>: Feeling or sensation of itchiness on your skin.

- Upper Airway Infection (like the common cold)
  - You may experience infections involving the nose, pharynx, larynx, and sinuses. Symptoms include a blocked (congested) nose, a runny nose, and sneezing. You may also have clear discharge (mucus) from the nose. You may feel generally unwell and may also be associated with fever. Treatment is usually supportive but if symptoms persist please inform your doctor
- Hand-Foot Syndrome (Plantar erythrodysaesthesia syndrome): When a small amount of drug leaks out of the blood vessels, it damages the surrounding tissues. Symptoms may include tingling, burning, redness, flaking, swelling, blistering, and sores of the hands and feet due to the increased friction and heat your extremities are exposed to. If you experience these symptoms, apply ice packs and elevate hands and feet, then contact your study doctor immediately for treatment.

#### Uncommon side effects: (Occurring in 0.1% up to less than 1% of patients):

- Myelodysplastic syndrome (MDS)<sup>a</sup> and acute myeloid leukemia (AML)<sup>a</sup> have been reported in a very small number of patients treated with rucaparib during the safety period (while on treatment with rucaparib and 28 days after last dose). MDS is a pre-cancerous condition where the bone marrow is not as good at producing blood cells (red and/or white blood cells and/or platelets). People with MDS need transfusions (red blood cells and/or platelets) and/or other treatments. In some cases, MDS can progress to AML, which is a cancer of the bone marrow where more abnormal and immature white blood cells (also called blasts) are made than normal white blood cells. People with AML need treatment with chemotherapy and/or a bone marrow transplant. Patients may develop AML without first being diagnosed with MDS.
- Events of MDS and AML have also been reported with PARP inhibitors similar to rucaparib. At this time it is not known whether rucaparib or other PARP inhibitors cause MDS or AML, or if these developed as a result of previous chemotherapy these patients received. Your study doctor will closely monitor your blood cell levels during treatment. If he/she has any concerns about your blood counts you may be asked to have a biopsy of your bone marrow.
  - <u>a</u>\_These risks have not yet been determined by Clovis as related to rucaparib. Some of these risks have been reported in a high frequency of patients in clinical trials involving rucaparib (e.g. itchy skin, rash), others have been reported in a small number of patients but pose significant risk (e.g. MDS/AML) or are generally known to be caused by other anti-cancer treatments (e.g. palmar-plantar erythrodysaesthesia).

The Study Doctor may decide to interrupt and/or reduce your rucaparib dose if you experience certain side effects. If your dose is reduced you will be given a new bottle of tablets.

There may be risks involved in taking this drug that have not yet been discovered. There is always a risk involved in taking an experimental drug but every precaution will be taken. If you suffer any side effects or injuries, or your condition gets worse, tell your study doctor immediately so you can receive appropriate care.

#### **Imaging Risks:**

This research study includes exposure to radiation from x-rays or gamma rays. This radiation exposure is for research purposes only and is not part of your medical care. X-rays and gamma rays from natural or medical sources can damage the genetic material (DNA) in your cells. At low doses, the body is usually able to repair the damage.

Date: March 31, 2022

Principal Investigator: Mark Markowski M.D. Ph.D.

Application No.: IRB00156514

The total radiation exposure may be up to 4.2 rem (a rem is a unit of absorbed radiation). The radiation exposure that you will get from screening CT guided biopsy is 0.8 rem. If you agree to the optional biopsy of your cancer and this is done by CT guided biopsy, you will receive an additional radiation exposure of 0.8 rem. You may receive an additional radiation exposure if you have one extra bone scan (0.8 rem) and one extra CT scan (1.8 rem) at the time of disease worsening (progression).

This is more than the 0.3 rem that the average person in the United States gets each year from natural sources like the sun, outer space, air, food and soil. It is less than the 5 rems of radiation that is allowed each year for people who are exposed to radiation in their jobs.

The radiation exposure described here is what you will get from this research study only. It does not include any exposure you may have received or will receive from other tests outside of this study that are a part of your medical care. Radiation risk builds up with each exposure. You should think about your own history of radiation exposure from tests (like x-rays or CT scans) in deciding about the radiation in this study. If you have questions about the total amount of radiation you will be receiving, you should ask your doctor.

#### Other Risks in the Study:

Your cancer may continue to grow if you elect to participate in this trial. You may develop symptoms from cancer or the cancer may spread during this clinical trial.

#### **Allergic Reactions**

As with any drug, it is possible that you could have allergic reactions to study drug, such as itching, skin rash, facial swelling, and/or a severe or sudden drop in blood pressure. A sudden drop in blood pressure could lead to shock with loss of consciousness and/or possible seizures, including the possibility of death. If you have any of the above symptoms, seek medical attention right away.

**Blood Draw:** Taking blood may cause discomfort, bleeding or bruising where the needle enters the body. In rare cases, it may result in fainting. There is a small risk of infection.

<u>Confidentiality:</u> There is the risk that information about you may become known to people outside this study.

Genetic information is unique to you and your family, even without your name or other identifiers. Johns Hopkins follows procedures to prevent people who work with your DNA information from being able to discover it belongs to you. However, new techniques are constantly being developed that may in the future make it easier to re-identify genetic data, so we cannot promise that your genetic information will never be linked to you.

There may be side effects and discomforts that are not yet known.

# 5. Are there risks related to pregnancy?

Rucaparib may cause harm to a fetus. Participants with partners capable of becoming pregnant who subsequently become pregnant may risk problems in the fetus. While taking the study drug, and for 4 months after stopping the study drug, you must use a condom when having sexual intercourse with a female partner, even if they are pregnant. Your female partner must also use a suitable method of contraception. Highly effective birth control is considered to be a method with a less than 1% per year failure rate and is defined in this study as established use of progesterone-only injectable or implantable contraceptives (e.g. Depo Provera, Implanon, Nexplanon), placement of an intrauterine device (IUD) or

Date: March 31, 2022

Principal Investigator: Mark Markowski M.D. Ph.D.

Application No.: IRB00156514

intrauterine system (IUS), surgical sterilization, or true, complete (as opposed to periodic) abstinence. If this applies to you, please discuss your plan for birth control with the investigator or study staff.

#### Transfer of Drug through Semen

Male patients must use a condom when having sex to avoid passing rucaparib to your partner through semen. You must also not make semen donations for 6 months following the last dose of rucaparib/study drug because rucaparib might damage sperm.

Tell your study doctor immediately if your partner becomes pregnant while taking you are on the study drug regimen or within 6 months for after your last dose of study drug. Please discuss with your doctor suitable methods of birth control.

This research may hurt an embryo or fetus in ways we do not currently know.

# 6. Are there benefits to being in the study?

You may or may not directly benefit from being in this study. If you take part in this study, you may help others in the future.

# 7. What are your options if you do not want to be in the study?

If you decide not to join this study, other options are available. You do not have to join this study to get treatment. Other treatments include androgen deprivation therapy with or without chemotherapy (Docetaxel) along with blood work, CT scans, and bone scans.

You do not have to join this study. If you do not join, your care at Johns Hopkins will not be affected.

# 8. Will it cost you anything to be in this study?

You will receive a separate Insurance and Research Participant Financial Responsibility Information Sheet (Sheet).

This Sheet will give you the following information:

- The procedures, tests, drugs or devices that are part of this research and that will be paid for by the study (no cost to you).
- The procedures, tests, drugs or devices that will be billed to you and/or your health insurer. If you have health insurance, you will be responsible for any co-pays or deductibles not covered by your insurance.

# 9. Will you be paid if you join this study?

You will not be paid to join this study.

# 10. Can you leave the study early?

- You can agree to be in the study now and change your mind later.
- If you wish to stop, please tell us right away.
- Leaving this study early will not stop you from getting regular medical care.

If you leave the study early, Johns Hopkins may use or give out your health information that it has already collected if the information is needed for this study or any follow-up activities.

Date: March 31, 2022

Principal Investigator: Mark Markowski M.D. Ph.D.

Application No.: IRB00156514

## 11. Why might we take you out of the study early?

You may be taken out of the study if:

- Staying in the study would be harmful.
- You need treatment not allowed in the study.
- You fail to follow instructions.
- The study is cancelled.
- There may be other reasons to take you out of the study that we do not know at this time.

If you are taken out of the study or stop taking the study drug, we will ask you to come in for a final visit about 1 month after your last dose of study drug. You will have a physical exam, blood tests, review of your medications, CT, and bone scan.

If you are taken out of the study early, Johns Hopkins may use or give out your health information that it has already collected if the information is needed for this study or any follow-up activities.

## 12. How will your privacy be protected?

We have rules to protect information about you. Federal and state laws and the federal medical Privacy Rule also protect your privacy. By signing this form you provide your permission, called your "authorization," for the use and disclosure of information protected by the Privacy Rule. The research team working on the study will collect information about you. This includes things learned from the procedures described in this consent form. They may also collect other information including your name, address, date of birth, and information from your medical records (which may include information about HIV status, drug, alcohol or STD treatment, genetic test results, or mental health treatment).

The research team who may be a part of Johns Hopkins Health System, Johns Hopkins University or the Johns Hopkins Applied Physics Laboratory will know your identity and that you are in the research study. Other people at Johns Hopkins, including your doctors, may also see or give out your information. We make this information available to your doctors for your safety.

People outside of Johns Hopkins may need to see or receive your information for this study. Examples include government agencies (such as the Food and Drug Administration), safety monitors, other sites in the study and companies that sponsor the study.

If you are in a cancer study that receives federal funding, the National Cancer Institute (NCI) now requires that we report identifiable information (such as, zip code) about your participation. You may contact the NCI if you have questions about how this information is used.

We cannot do this study without your authorization to use and give out your information. You do not have to give us this authorization. If you do not, then you may not join this study.

We will use and disclose your information only as described in this form and in our Notice of Privacy Practices; however, people outside Johns Hopkins who receive your information may not be covered by this promise or by the federal Privacy Rule. We try to make sure that everyone who needs to see your information keeps it confidential – but we cannot guarantee that your information will not be redisclosed.

Date: March 31, 2022

Principal Investigator: Mark Markowski M.D. Ph.D.

Application No.: IRB00156514

The use and disclosure of your information has no time limit. You may revoke (cancel) your permission to use and disclose your information at any time by notifying the Principal Investigator of this study by phone or in writing. If you contact the Principal Investigator by phone, you must follow-up with a written request that includes the study number and your contact information. The Principal Investigator's name, address, phone and fax information are on page one of this consent form.

If you do cancel your authorization to use and disclose your information, your part in this study will end and no further information about you will be collected. Your revocation (cancellation) would not affect information already collected in the study, or information we disclosed before you wrote to the Principal Investigator to cancel your authorization.

# 13. Will the study require any of your other health care providers to share your health information with the researchers of this study?

As a part of this study, the researchers may ask to see your health care records from your other health care providers.

# 14. What treatment costs will be paid if you are injured in this study?

Johns Hopkins does not have a program to pay you if you are hurt or have other bad results from being in the study. However, medical care at Johns Hopkins is open to you as it is to all sick or injured people.

The costs for any treatment or hospital care you receive as the result of a study-related injury that are not covered by a health insurer will be billed to you.

By signing this form you will not give up any rights you have to seek compensation for injury.

# 15. What other things should you know about this research study?

a. What is the Institutional Review Board (IRB) and how does it protect you?

The Johns Hopkins Medicine IRB is made up of:

- Doctors
- Nurses
- Ethicists
- Non-scientists
- and people from the local community.

The IRB reviews human research studies. It protects the rights and welfare of the people taking part in those studies. You may contact the IRB if you have questions about your rights as a participant or if you think you have not been treated fairly. The IRB office number is 410-955-3008. You may also call this number for other questions, concerns or complaints about the research.

When the Johns Hopkins School of Medicine Institutional Review Board (IRB) reviews a study at another site, that site (institution) is solely responsible for the safe conduct of the study and for following the protocol approved by the Johns Hopkins IRB.

#### b. What do you do if you have questions about the study?

Call the principal investigator, Dr. Mark C. Markowski at 410-955-8893. If you wish, you may contact the principal investigator by letter or by fax. The address and fax number are on page one of this consent form. If you cannot reach the principal investigator or wish to talk to someone else, call the IRB office at 410-955-3008.

Date: March 31, 2022

Principal Investigator: Mark Markowski M.D. Ph.D.

Application No.: IRB00156514

#### c. What should you do if you are injured or ill as a result of being in this study?

If you think you are injured or ill because of this study, call Dr. Mark C. Markowski at 410-955-8893 during regular office hours.

**If you have an urgent medical problem** related to your taking part in this study, call the medical oncology clinic at 410-955-8893 during regular office hours and at 410-955-4331 after hours and on weekends.

#### d. What happens to Data and Biospecimens that are collected in the study?

Johns Hopkins and our research partners work to understand and cure diseases. The biospecimens and/or data you provide are important to this effort.

If you join this study, you should understand that you will not own your biospecimens or data, and should researchers use them to create a new product or idea, you will not benefit financially.

With appropriate protections for privacy, Johns Hopkins may share your biospecimens and information with our research sponsors and partners.

Date: March 31, 2022

Principal Investigator: Mark Markowski M.D. Ph.D.

Application No.: IRB00156514

# 16. What does your signature on this consent form mean?

Your signature on this form means that: You understand the information given to you in this form, you accept the provisions in the form and you agree to join the study. You will not give up any legal rights by signing this consent form.

#### WE WILL GIVE YOU A COPY OF THIS SIGNED AND DATED CONSENT FORM

| Signature of Participant | (Print Name) | Date/Time |
|---|---|---|
| Signature of Person Obtaining Consent | (Print Name) | Date/Time |
| - g | () | |
| Signature of Witness to Consent Procedures<br>(optional unless IRB or Sponsor required) | (Print Name) | Date/Time |
| I have received the separate Insurance and Research | n Participant Financial Responsibility In | formation Sheet. |
| Signature of Participant, LAR or Parent/Guardian | (Print Name) | Date/Time |
| 2.5 Of I dividipant, Diffe of I divid Oddidimi | (Time Tame) | Dute, Time |

NOTE: A COPY OF THE SIGNED, DATED CONSENT FORM MUST BE KEPT BY THE PRINCIPAL INVESTIGATOR AND A COPY MUST BE GIVEN TO THE PARTICIPANT. IF APPROPRIATE FOR THIS STUDY, A SCANNED COPY OF THE SIGNED CONSENT FORM SHOULD BE UPLOADED TO THE PARTICIPANT'S EPIC/EMR RECORD (UNLESS NO MEDICAL RECORD EXISTS OR WILL BE CREATED).

Date: March 31, 2022

Principal Investigator: Mark Markowski M.D. Ph.D.

Application No.: IRB00156514

# DOCUMENTATION OF PHYSICIAN/MID-LEVEL PROVIDER CONSENT PROCESS

| My signature below indicates that I have discussed the risks, benefits, and alternatives, answered any questions, and believe the participant is able to make an informed choice to join the study. | | |
|---|---|---|
| nature of Physician/Mid-Level Provider | (Print Name) | Date/Time |
| CD (iii | | Date/Time |
| nature of Participant | (Print Name) | Date/11me |
| nature of Witness to Consent Procedures<br>tional unless IRB or Sponsor required) | (Print Name) | Date/Time |
| UST BE GIVEN TO THE PARTICIPANT. | CONSENT FORM MUST BE KEPT BY THE PRINC<br>IF APPROPRIATE FOR THIS STUDY, A SCANNE<br>ARTICIPANT'S EPIC/EMR RECORD (UNLESS N | ED COPY OF THE SIGNED CONSE |
| , | | |